CLINICAL TRIAL: NCT02630628
Title: A Randomized Open-label Study to Evaluate the Efficacy and Safety of Tacrolimus and Corticosteroids in Comparison With Mycophenolate Mofetil and Corticosteroids in Subjects With Class III/IV±V Lupus Nephritis
Brief Title: Efficacy and Safety of Tacrolimus Versus Mycophenolate in Lupus Nephritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Daniel Tak-Mao Chan, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALNN-IIS-17JUL15-1
Record Dates: First submitted 2015-12-05; First posted 2015-12-15 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis; mycophenolate mofetil; tacrolimus
MeSH Terms: conditions — Lupus Nephritis | interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus (Experimental): route: oral duration: 96 weeks
  Interventions: Drug: Tacrolimus
- Mycophenolate Mofetil (Active Comparator): route: oral duration: 96 weeks
  Interventions: Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Tacrolimus — Dosage: start at 2mg twice a day, then titrated according to therapeutic drug level monitoring using 12-hour post-dose blood sampling
  Other Names: Prograf
  Arms: Tacrolimus
Drug: Mycophenolate mofetil — Dosage: start at 1g twice a day, then taper as per protocol
  Other Names: Cellcept
  Arms: Mycophenolate Mofetil

SUMMARY:
Prospective, randomized, parallel-group controlled, open-label, international (Asian) multicenter, comparison of corticosteroids combined with tacrolimus and corticosteroids combined with mycophenolate mofetil.

DETAILED DESCRIPTION:
There is accumulating evidence that tacrolimus (TAC) could serve as an effective medication for the treatment of lupus nephritis (LN). TAC is a calcineurin inhibitor, which is a key component in first-line combination immunosuppressive regimens after kidney transplantation, based on its proven efficacy in the prevention and treatment of allograft rejection and acceptable tolerability profile. Although it primarily targets T lymphocyte activation, its immunosuppressive actions encompass multiple immune response pathways due to the complex interactions between different cellular and soluble immune mediators. Moreover, the effect of calcineurin inhibitors on podocyte morphology and function, independent of their immunosuppressive effect, has translated into therapeutic efficacy in the treatment of proteinuric glomerular diseases such as membranous nephropathy and focal segmental glomerulosclerosis. Recent data from short-term studies showed that combination immunosuppressive regimens that included TAC and corticosteroids with or without mycophenolate mofetil (MMF) appeared at least as effective as other standard-of-care treatments for Class III/IV±V LN, and the inclusion of TAC might lead to more effective suppression of proteinuria. There is also preliminary data on its favorable tolerability when used as long-term maintenance treatment. This study aims to examine the role of TAC combined with corticosteroids, in comparison with the most commonly used standard-of-care treatment MMF plus corticosteroids, in the management of lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven LN Class III/IV±V (ISN/RPS 2003), with biopsy performed within 12 weeks of randomization.
2. Positive anti-dsDNA.
3. Active LN with proteinuria (urine protein/creatinine ratio ≥1.0 or 24-hr urine protein ≥1.0 g at baseline), with or without hematuria.
4. Both 'incident' (i.e. new) patients and 'flare' patients can be included.
5. Males or females aged 18 to 75 years inclusive at the time of screening.

Exclusion Criteria:

1. Renal disease unrelated to SLE (e.g. diabetes mellitus, other glomerular or tubulointerstitial disease, renovascular disease), or transplanted kidney.
2. Estimated glomerular filtration rate (eGFR by MDRD) ≤20 mL/min per 1.73 m2 or serum creatinine ≥300 micromol/L (3.39 mg/dL) at screening.
3. Renal biopsy showing cellular or fibrocellular crescent in more than 25% of glomeruli.
4. CNS or other severe organ manifestation of lupus that necessitate aggressive immunosuppressive therapy on its own.
5. Co-morbidities that require corticosteroid therapy (e.g. asthma, inflammatory bowel disease).
6. Treatment with prednisolone (or prednisone, or equivalent) at ≥20 mg/D for over 4 weeks within the past 3 months.
7. Treatment with MMF at >1.5 g/D for over 4 weeks within the past 3 months.
8. Known hypersensitivity or intolerability to prednisolone (or prednisone, or equivalent), TAC, or MMF at a dose of 1.25 g or below per day.
9. Subjects who are already on treatment with TAC, cyclosporine or any other calcineurin inhibitor on the day of screening; or have received treatment with TAC, cyclosporine or other calcineurin inhibitor for over 4 weeks within the past 6 months.
10. Treatment with cyclophosphamide, leflunomide, or methotrexate for over 2 weeks, or use of biological agent(s) regardless of duration, within the past 6 months (Note: prior use of azathioprine, mizoribine, intravenous immunoglobulins and anti-malarials is allowed).
11. Uncontrolled hypertension with systolic BP >160 mmHg or diastolic BP >95 mmHg.
12. Women who are pregnant or breastfeeding.
13. Women with childbearing potential or their male partners, who refuse to use an effective birth control method

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-12-05 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Efficacy of combined corticosteroids and TAC compared to combined corticosteroids and MMF in achieving sustained renal response (RR) in patients with active lupus nephritis [Class III/IV±V (LN)] | 96 weeks
  Sustained RR defined as satisfying all of the following criteria:
  1. proteinuria improved by ≥50% compared with baseline
  2. 24-hr urine protein <1 g
  3. serum creatinine not higher than 15% above baseline level or eGFR not less than 60 mL/min/1.73m2
  4. no occurrence of disease flare AFTER achieving response to treatment. Disease flare is defined as the need for 'rescue' immunosuppressive therapy with any one of the following i. increase of prednisolone dose from ≤7.5 mg/D to ≥15 mg/D for 4 weeks or longer ii. change of originally assigned immunosuppressive agent iii. addition of immunosuppressive medications prohibited in protocol

SECONDARY OUTCOMES:
Rate of complete renal remission | 96 weeks
  * proteinuria not higher than 0.5 g/D
  * serum creatinine not higher than 15% above baseline level or eGFR not less than 60 mL/min/1.73m2
Rate of partial renal remission | 96 weeks
  * proteinuria above 0.5 g/D and below 3 g/D and with ≥50% improvement compared with baseline level
  * serum creatinine not higher than 15% above baseline level or eGFR not less than 60 mL/min/1.73m2
Efficacy of combined corticosteroids and TAC compared to combined corticosteroids and MMF in achieving sustained renal response (RR) in patients with active lupus nephritis [Class III/IV±V (LN)] | 48 weeks
  Sustained RR defined as satisfying all of the following criteria:
  1. proteinuria improved by ≥50% compared with baseline
  2. 24-hr urine protein <1 g
  3. serum creatinine not higher than 15% above baseline level or eGFR not less than 60 mL/min/1.73m2
  4. no occurrence of disease flare AFTER achieving response to treatment. Disease flare is defined as the need for 'rescue' immunosuppressive therapy with any one of the following i. increase of prednisolone dose from ≤7.5 mg/D to ≥15 mg/D for 4 weeks or longer ii. change of originally assigned immunosuppressive agent iii. addition of immunosuppressive medications prohibited in protocol
Refractory disease | 96 weeks
  Never achieving partial renal remission since commencement of study
Rate of non-renal flare | 96 weeks
  Disease flare defined by the need for 'rescue' immunosuppressive therapy with any one of the following i. increase of prednisolone dose from ≤7.5 mg/D to ≥15 mg/D for 4 weeks or longer ii. change of originally assigned immunosuppressive agent iii. addition of immunosuppressive medications prohibited in protocol
Incidence of acute kidney injury | 96 weeks
  Number of patients who had increase of serum creatinine level ≥15% from baseline and whether the increase was reversible or irreversible
Incidence of TAC blood level above target range | 96 weeks
  Number of patients who had 12-hour post dose TAC blood level above i. 8 ng/mL (from baseline to end of week 24) ii. 7 ng/mL (from start of week 25 to end of week 48, and from start of week 49 to end of week 96 for patients who had serum creatinine level <150 micromol/L) iii. 6 ng/mL (from start of week 49 to end of week 96 for patients who had serum creatinine level ≥150 micromol/L)
Incidence of new onset hypertension or worsening hypertensive control | 96 weeks
  Number of patients who had new onset hypertension (blood pressure >140/90 mmHg) or worsening hypertensive control that required increase of number or dose of anti-hypertensive medications
Rate of infection | 96 weeks
  Number of patients who had infection that required hospitalization and its causative agents
Rate of Hospitalization | 96 weeks
  Number of patients who had been hospitalized, the cause and duration of hospitalization
Incidence of hyperkalemia | 96 weeks
  Number of patients who had serum potassium level >5.6 mmol/L
Incidence of metabolic acidosis | 96 weeks
  Number of patients who had serum bicarbonate level <17 mmol/L
Incidence of new onset diabetes mellitus | 96 weeks
  Number of patients who had fasting glucose > 6.0 mmol/L and/or required addition of blood glucose lowering drug(s)
Incidence of new onset hypercholesterolemia | 96 weeks
  Number of patients who had total cholesterol> 5.0 mmol/L and low density lipoprotein >3.4 mmol/L presented at 6 months or beyond from baseline and/or required addition of lipid-lowering drug(s)
Rate of treatment intolerance leading to premature study discontinuation | 96 weeks
  Definition of treatment intolerance i. severe gastrointestinal disturbance or marrow suppression (white blood cell count <2×10^9/L OR platelet count <50×10^9/L OR hemoglobin <8 g/dL) judged due to MMF and persisted despite reduction of MMF dosage to < 1.25 g per day ii. significant hand-tremor or neurotoxicity related to TAC
Rate of disease complication leading to premature study discontinuation | 96 weeks
  Number of patients who developed complication that led to premature study discontinuation
Rate of disease flare leading to premature study discontinuation | 96 weeks
  Disease flare is defined as the need for 'rescue' immunosuppressive therapy with any one of the following i. increase of prednisolone dose from ≤7.5 mg/D to ≥15 mg/D for 4 weeks or longer ii. change of originally assigned immunosuppressive agent iii. addition of immunosuppressive medications prohibited in protocol
Number of patients who failed to adhere to protocol defined corticosteroid reduction regimen | 96 weeks
  Failure to adhere to corticosteroid reduction regimen was defined as deviation from protocol-defined corticosteroid dose by >5mg/D for >3 weeks due to unsatisfactory treatment response or new-onset disease activity.
Incidence of adverse events | 96 weeks
  Number and type of adverse events, irrespective of whether the event was treatment-related or not
Incidence of serious adverse events | 96 weeks
  Number and type of serious adverse events, irrespective of whether the event was treatment-related or not
Changes in SELENA-SLEDAI scores | 96 weeks
  Changes in SELENA-SLEDAI scores from baseline to week 96
Changes in PGA scores | 96 weeks
  Changes in PGA scores from baseline to week 96
Changes in SFI scores | 96 weeks
  Changes in SFI scores from baseline to week 96
Changes in BILAG (2004) scores | 96 weeks
  Changes in BILAG (2004) scores from baseline to week 96

CONTACTS AND LOCATIONS:
Overall Officials: Tak-Mao Daniel Chan, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No